CLINICAL TRIAL: NCT00157807
Title: Clinical and Economic Consequences of Left Atrial Bipolar Radiofrequency Ablation of Persistent and Permanent Atrial Fibrillation During Cardiac Surgery. A Prospective Randomized Multi Center Trial
Brief Title: Clinical and Economic Consequences of Left Atrial Bipolar Radiofrequency Ablation of Persistent and Permanent Atrial Fibrillation During Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no eligible patients can be found
Sponsor: Medtronic Cardiac Surgery (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CEN_G_CS_1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
Keywords: Persistent Atrial Fibrillation; Permanent Atrial Fibrillation; Mitral Valve Defect; Tricuspid Valve Defect; Aortic Valve Defect
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Ablation (No Intervention)
- bipolar radiofrequency ablation of persistent and permanent AF (Other): intra operative bipolar RF ablation of persistent and permanent AF
  Interventions: Procedure: bipolar radiofrequency ablation of persistent and permanent AF

INTERVENTIONS:
Procedure: bipolar radiofrequency ablation of persistent and permanent AF
  Arms: bipolar radiofrequency ablation of persistent and permanent AF

SUMMARY:
The clinical effects of intra-operative radiofrequency ablation in patients with persistent or permanent atrial fibrillation and an indication for an implantation of a heart valve prosthesis or coronary bypass surgery are the purposes of this study. The study will examine if and to what extent the quality of life and the use of medical care differs between patients with and without ablation. Furthermore, there will be thorough echocardiographic examinations of the heart to detect differences between the different treatment groups. The patients will be followed for one year after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation
* Permanent atrial fibrillation
* Mitral valve defect
* Tricuspid valve defect
* Aortic valve defect
* Coronary artery disease

Exclusion Criteria:

* Pregnancy
* Age < 18 or > 75 Years
* Emergency surgery
* Left dominant coronary circulation (relative contraindication)
* Coronary arteries of the posterior wall without pathological findings: No inclusion
* Stenosis of the posterior wall vessels, supplied with a CABG (coronary artery bypass grafting): Inclusion possible
* Left ventricular ejection fraction < 30%
* Size of the left atrium > 7 cm
* Thrombosis of the left atrial appendage
* Leads in the coronary sinus
* Atrial flutter
* Infective endocarditis
* Reoperation
* Participation in other studies
* Life expectancy of less than 12 months
* Psychiatric disorders
* Hyperthyreosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Quality of life | 12 months
Cost of care | 12 months

SECONDARY OUTCOMES:
Atrial fibrillation | 12 months
Echo parameters | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Calin Vicol, Professor, Principal Investigator — Klinikum der Universität München Großhadern Cardiac Surgery
Locations (5):
- Germany (5):
  - Klinik für Herz-, Thorax- und Gefäßchirurgie, Lahr, Baden-Wurttemberg
  - Klinikum der Universität Muenchen Großhadern Cardiac Surgery, München, Bavaria
  - Klinik für Herz- und Thoraxchirurgie, Bochum, North Rhine-Westphalia
  - Klinik und Poliklinik für Herzchirurgie der Rhein. Friedrich-Wilhelms-Universität Bonn, Bonn, North Rhine-Westphalia
  - Klinik für Herz- und Thoraxchirurgie der Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony

REFERENCES:
- See also: Klinikum der Universität — http://www.klinikum.uni-muenchen.de
- See also: Herzchirurgie — http://hch.klinikum.uni-muenchen.de